CLINICAL TRIAL: NCT00002052
Title: Prospective Comparison of Ampicillin / Amoxicillin Versus Ceftriaxone for the Treatment of Salmonella Infections in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 019A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: HIV Infections; Salmonella Infections
Keywords: Salmonella Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Amoxicillin; Ceftriaxone
MeSH Terms: conditions — HIV Infections; Salmonella Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Ceftriaxone; Ampicillin; Amoxicillin

INTERVENTIONS:
Drug: Ceftriaxone sodium
Drug: Ampicillin sodium
Drug: Amoxicillin trihydrate

SUMMARY:
To compare the effectiveness of standard treatment with parenteral ampicillin and oral amoxicillin compared to initial daily therapy with ceftriaxone followed by 3 times weekly suppressive treatment for salmonella infections in AIDS patients.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Type I hypersensitivity to beta-lactam antibiotics.
* Not expected to survive 12 weeks.
* In a coma or with other central nervous system (CNS) impairment.

Patients with the following are excluded:

* Type I hypersensitivity to beta-lactam antibiotics.
* Not expected to survive 12 weeks.
* In a coma or with other central nervous system (CNS) impairment.

Prior Medication:

Excluded within 48 hours of study entry:

* Treatment with an antibiotic active in vitro against Salmonella.

HIV infection, AIDS, or AIDS related complex (ARC).

* Salmonella bacteremia or positive stool culture in patient with 3 or more stools per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County - USC Med Ctr, Los Angeles, California, United States